CLINICAL TRIAL: NCT01939301
Title: Randomized Trial of Inhaled Nitric Oxide to Treat Acute Pulmonary Embolism
Brief Title: Nitric Oxide to Treat Pulmonary Embolism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Collaborators: Mallinckrodt (Industry); National Institutes of Health (NIH) (NIH); University of Mississippi Medical Center (Other); University of Texas, Southwestern Medical Center at Dallas (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jeffrey Kline, Vice Chair of Research, Indiana University School of Medicine
Organization: Indiana University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Kline-1UM NO for PE; 1UM1HL113203-01A1 (NIH)
Record Dates: First submitted 2013-08-28; First posted 2013-09-11 (Estimated); Results first posted 2018-03-29 (Actual); Last update posted 2018-10-03 (Actual); Status verified 2018-09

CONDITIONS: Pulmonary Embolism
Keywords: Pulmonary embolism clot
MeSH Terms: conditions — Pulmonary Embolism | interventions — salicylhydroxamic acid; Oxygen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inhaled Nitric Oxide (Active Comparator): Inhaled nitric oxide
  Interventions: Drug: Inhaled Nitric Oxide
- Placebo (Placebo Comparator): Oxygen
  Interventions: Drug: Sham

INTERVENTIONS:
Drug: Inhaled Nitric Oxide — Nitric Oxide + oxygen
  Arms: Inhaled Nitric Oxide
Drug: Sham — Nitrogen + Oxygen
  Other Names: placebo; oxygen
  Arms: Placebo

SUMMARY:
This is a randomized study to treat subjects diagnosed with pulmonary embolism with inhaled nitric oxide or placebo (oxygen).

DETAILED DESCRIPTION:
This is a randomized, double blind study to treat subjects diagnosed with pulmonary embolism with inhaled nitrix oxide. In this clinical trial investigators will randomized patients to receive inhaled nitric oxide or sham (nitrogen + oxygen) for 24 hours. Patients must have a submassive pulmonary embolism (PE) and evidence of right ventricular (RV) heart dysfunction. Investigators hypothesize that the administration of inhaled NO + oxygen to patients with severe submassive PE will improve RV function, reduce RV strain and necrosis and improve dyspnea (difficulty breathing) more than sham oxygen treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18
* Pulmonary imaging-proven PE, as interpreted by local radiologist
* At least one predictor of RV dysfunction:

  1. echocardiography with RV dilation or hypokinesis,
  2. estimated RVSP >40mm HG,
  3. RV>LV on CTPA,
  4. elevated troponin I (>0.1 ng/mL) or natriuretic peptide (BNP > 90 pg/mL),
  5. screening bedside cardiac ultrasound with color flow capability that shows RV dysfunction,
  6. RV strain on ECG
* Plan to admit to a bed with telemetry capability

Exclusion Criteria:

* Vasopressor support at time of enrollment
* Pregnancy
* Plan by clinical care team to use lytic or surgical embolectomy
* Plan by clinical team to use platelet inhibiting drugs
* Contraindication to anticoagulation
* Altered mental status such that the patient is unable to provide informed consent
* Inability to use a nasal cannula or face mask
* Comfort care measures instituted
* Supplemental oxygen requirements greater than can be administered via nasal cannula in order to maintain Sa)2 > 80%
* Pneumothorax with decompression
* Serum MetHb > 10%
* Recent use of drugs known to increase cGMP
* Use of nitroprusside or nitroglycerin within the last 4 hours
* Use of any other nitrates with in the past 24 hours
* Use of a fibrinolytic medicine within the past 14 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2013-10; Primary Completion 2016-10-31 (Actual); Study Completion 2016-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff A Kline, MD, Principal Investigator — Indiana University
Locations (4):
- United States (4):
  - Eskenazi Hospital, Indianapolis, Indiana
  - Indiana University Hospital, Indianapolis, Indiana
  - Methodist Hospital, Indianapolis, Indiana
  - University of Mississippi, Jackson, Mississippi

REFERENCES:
- [Derived] Kline JA, Puskarich MA, Jones AE, Mastouri RA, Hall CL, Perkins A, Gundert EE, Lahm T. Inhaled nitric oxide to treat intermediate risk pulmonary embolism: A multicenter randomized controlled trial. Nitric Oxide. 2019 Mar 1;84:60-68. doi: 10.1016/j.niox.2019.01.006. Epub 2019 Jan 8. PMID 30633959
- [Derived] Kline JA, Hall CL, Jones AE, Puskarich MA, Mastouri RA, Lahm T. Randomized trial of inhaled nitric oxide to treat acute pulmonary embolism: The iNOPE trial. Am Heart J. 2017 Apr;186:100-110. doi: 10.1016/j.ahj.2017.01.011. Epub 2017 Jan 27. PMID 28454823

RESULTS

PARTICIPANT FLOW:
Groups:
- Sham: oxygen
  Nitrogen + Oxygen
Period: Overall Study
Arm/Group | Inhaled Nitric Oxide | Sham
Started | 39 | 39
Completed | 38 | 38
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inhaled Nitric Oxide | Sham | Total
Number analyzed (Participants) | 39 | 39 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (15) | 59 (16) | 57 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 20 | 41
  Male | 18 | 19 | 37
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 39 | 39 | 78

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Normal Right Ventricular (RV) Function and Viability
Description: Right ventricular (RV) function and viability assessed by the composite of normal RV size (<42 mm in diastole) and tricuspid annular plane systolic excursion (TAPSE) > 16 mm and normal right ventricular index of myocardial performance (RIMP) < 0.40 using spectral Doppler or < 0.55 using tissue Doppler) and normal fractional area change (FAC) (> 33%) and a serum hsTnT < 14pg/mL. Missing values will be considered normal.
Time Frame: 5 days or hospital discharge (whichever occurs first)
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Nitric Oxide | Sham
Number analyzed (Participants) | 38 | 38
Participants | 9 | 5

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Inhaled Nitric Oxide | Sham
All-Cause Mortality (participants affected / at risk) | 2/38 | 2/38
Serious Adverse Events (participants affected / at risk) | 2/38 | 2/38
Other Adverse Events (participants affected / at risk) | 12/38 | 11/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inhaled Nitric Oxide (N=38) | Sham (N=38)
death (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inhaled Nitric Oxide (N=38) | Sham (N=38)
arrhythmia (Cardiac disorders) | 12 (12) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes